CLINICAL TRIAL: NCT03428152
Title: The Efficacy of Superior Hypogastric Blockade for Postoperative Pain
Brief Title: Superior Hypogastric Blockade for Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hande Gurbuz, M.D., Principal investigator, Derince Training and Research Hospital
Other Study IDs: U1111-1205-2226
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Results first posted 2019-06-03 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Superior Hypogastric Plexus Block; Hysterectomy; Pain, Postoperative; Gynecologic Disease
Keywords: superior hypogastric plexus block; hysterectomy; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypo: The participants with a superior hypogastric block
  Interventions: Procedure: superior hypogastric block
- NoHypo: The participants without a superior hypogastric block; the patients with an epidural catheter, who receive a different block technique (ie: TAP block), or who are unsuitable for SHP block (ie: if retro-peritoneum is opened intraoperatively by the surgeon)

INTERVENTIONS:
Procedure: superior hypogastric block — superior hypogastric blockade during surgery
  Groups: Hypo

SUMMARY:
The primary indication for superior hypogastric (SHP) block is visceral pelvic pain, most commonly from malignancy of the ovary, uterus, cervix, bladder, rectum or prostate. Percutaneous SHP blocks should be done under guidance of ultrasonography, fluoroscopy, magnetic resonance or computed tomography. Because of the close proximity of SHP to major vessels, and structures like vertebral column (for posterior) and guts (for anterior) are being on the way of the needle, these percutaneous blocks are associated with serious complications. Performing SHP during hysterectomy surgery, gives advantages to rule out these complications by exploring the whole intraabdominal anatomy.

The investigators' theory is to find out if SHP blocks (during pelvic surgery) are useful for decreasing VAS pain scores and opioid consumption for postoperative pain.

DETAILED DESCRIPTION:
Nerve blocks are frequently used in daily practice as an anesthetic and analgesia technique for surgery, postoperative pain and chronic pain. Total abdominal hysterectomy causes significant postoperative pain. Epidural blocks are frequently preferred for postoperative pain control, since most of the anesthetists are skilled with neuraxial blocks. However, an epidural catheter placement and epidural injections have some side effects and complications.

Pelvis is innervated by thoracolumbar and sacral segments. Autonomic (sympathetic and parasympathetic) and somatic (motor and sensory) nerves provide innervation of pelvis. The sympathetic nervous system, which transmits nociceptive messages from the viscera to brain, plays an important role in the transmission of visceral pain. Generally, in order to block transmission of nociceptive information from the pelvic viscera to the spinal cord, interruption of sympathetic pathways will be necessary. The sympathetic nerve block on the sympathetic nervous system for the management of chronic pelvic pain has been proposed at three main levels: ganglion impar, hypogastric plexus and L2 lumbar sympathetic blocks. By following the pelvic anatomy, there could be an alternative way for acute pain relief for abdominal hysterectomy: superior hypogastric block.

The superior hypogastric plexus lies retroperitoneally in front of L4 as a bunch of fibers. As these fibers descend, at the level of L5 they divide into the hypogastric nerves. The hypogastric nerves pass downward from L5-S1, following the concave curve of the sacrum and passing on each side of the rectum to form the inferior hypogastric plexus. These nerves continue their down¬ward course along each side of the bladder to provide innervation to the pelvic viscera and vasculature.

The primary indication for superior hypogastric block (SHNB) is visceral pelvic pain, most commonly from malignancy of the ovary, uterus, cervix, bladder, rectum or prostate. Percutaneous SHP blocks can be done by using posterior approach (transdiscal) and paravertebral) and anterior techniques. All of these interventions should be done under guidance of ultrasonography, fluoroscopy, magnetic resonance or computed tomography. Because of the close proximity of SHP to major vessels, and structures like vertebral column (for posterior) and guts (for anterior) are being on the way of the needle, these percutaneous blocks are associated with complications.

SHP block has been performed by anesthetists or surgeons in Kocaeli Derince Training and Research Hospital regularly since they have discovered the advantages of this block technique. Performing SHP block during hysterectomy surgery, gives advantages to rule out these complications by exploring the whole intraabdominal anatomy. Based on the complexity of the pelvic innervation, SHP blocks do not offer a total painless period like central neuraxial blocks for sure. If SHP block is performed in patients who do not have epidural catheters, it can be useful to decrease postoperative pain scores and opioid or NSAID consumption significantly.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II
* Elective hysterectomy

Exclusion Criteria:

* ASA III
* Different kind of surgery
* Known allergy to local anesthetic drugs
* Different analgesia protocol (ie: epidural, TAP block,..)
* Refusal of the patient

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients who are scheduled for hysterectomy
Study Population: The patients who are scheduled for elective hysterectomy under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hande G. Aytuluk, MD, Principal Investigator — Derince Training and Research Hospital; Gulfem Basol, MD, Study Chair — Derince Training and Research Hospital; Ahmet Kale, Prof, Study Chair — Derince Training and Research Hospital; Canan Balci, Assoc Prof, Study Chair — Derince Training and Research Hospital
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators do not prefer to share the study plan and records.

REFERENCES:
- [Background] Plancarte R, de Leon-Casasola OA, El-Helaly M, Allende S, Lema MJ. Neurolytic superior hypogastric plexus block for chronic pelvic pain associated with cancer. Reg Anesth. 1997 Nov-Dec;22(6):562-8. PMID 9425974
- [Background] de Leon-Casasola OA, Kent E, Lema MJ. Neurolytic superior hypogastric plexus block for chronic pelvic pain associated with cancer. Pain. 1993 Aug;54(2):145-151. doi: 10.1016/0304-3959(93)90202-Z. PMID 8233527
- [Background] Sindt JE, Brogan SE. Interventional Treatments of Cancer Pain. Anesthesiol Clin. 2016 Jun;34(2):317-39. doi: 10.1016/j.anclin.2016.01.004. PMID 27208713
- [Background] Choi JW, Kim WH, Lee CJ, Sim WS, Park S, Chae HB. The Optimal Approach for a Superior Hypogastric Plexus Block. Pain Pract. 2018 Mar;18(3):314-321. doi: 10.1111/papr.12603. Epub 2017 Jul 6. PMID 28520297
- [Background] Turker G, Basagan-Mogol E, Gurbet A, Ozturk C, Uckunkaya N, Sahin S. A new technique for superior hypogastric plexus block: the posteromedian transdiscal approach. Tohoku J Exp Med. 2005 Jul;206(3):277-81. doi: 10.1620/tjem.206.277. PMID 15942158
- [Background] Erdine S, Yucel A, Celik M, Talu GK. Transdiscal approach for hypogastric plexus block. Reg Anesth Pain Med. 2003 Jul-Aug;28(4):304-8. doi: 10.1016/s1098-7339(03)00191-3. PMID 12945023
- [Result] Rapp H, Ledin Eriksson S, Smith P. Superior hypogastric plexus block as a new method of pain relief after abdominal hysterectomy: double-blind, randomised clinical trial of efficacy. BJOG. 2017 Jan;124(2):270-276. doi: 10.1111/1471-0528.14119. Epub 2016 Jun 12. PMID 27292167
- [Derived] Aytuluk HG, Kale A, Astepe BS, Basol G, Balci C, Colak T. Superior Hypogastric Plexus Blocks for Postoperative Pain Management in Abdominal Hysterectomies. Clin J Pain. 2020 Jan;36(1):41-46. doi: 10.1097/AJP.0000000000000767. PMID 31567396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypo | NoHypo
Started | 37 | 41
Completed | 30 | 30 (exclusions: epidural / TAP / wound infiltration malignity retroperitone was opened age >65)
Not Completed | 7 | 11
Not completed — Physician Decision | 4 | 2
Not completed — Protocol Violation | 3 | 5
Not completed — Lack of Efficacy | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypo | NoHypo | Total
Number analyzed (Participants) | 37 | 41 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.36 (6.51) | 51.63 (7.49) | 52 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 78
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 37 | 41 | 78

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Scores
Description: Patients' pain scores will be scored with a 10 cm Visual Analogue Scale (VAS). Each will be scored between 0-10 (0: no pain; 10: worst pain ever) (PACU: Post-anesthesia care unit) VAS-PACU: VAS scores at PACU VAS 1: VAS scores at postoperative 1st hour (ward) VAS 6: VAS scores at postoperative 6th hour (ward) VAS 12: VAS scores at postoperative 12th hour (ward) VAS 24: VAS scores at postoperative 24th hour (ward) VAS 48: VAS scores at postoperative 48th hour (ward)
Time Frame: postoperative 48 hour follow-up (PACU and ward)
Population: 37 patients with a superior hypogastric block (7 was excluded); 41 patients without a superior hypogastric block (11 was excluded).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypo | NoHypo
Number analyzed (Participants) | 37 | 41
units on a scale
  VAS PACU | 4.76 (1.55) | 7.38 (1.63)
  VAS 1 | 3.7 (3.36) | 6.66 (2.10)
  VAS 6 | 1.9 (1.32) | 4.23 (2.03)
  VAS 12 | 0.83 (0.74) | 3.16 (2.13)
  VAS 24 | 0.53 (0.68) | 2.1 (2.17)
  VAS 48 | 0.2 (0.4) | 1.2 (1.39)

2. Primary Outcome: Postoperative Analgesic Consumption
Description: Total number of non-steroid anti-inflammatory drug (NSAID) and opioid vials that are applied to patients in post-anesthesia care unit (PACU) and at ward will be recorded.
  Target VAS score for NSAID is >4; if there is no response to NSAID and pain is worsening opioid drugs will be applied (this is our routine clinical practice) NSAID: Diclofenac sodium 75mg per vial; opioid: Tramadol 100mg per vial.
Time Frame: postoperative 48 hour follow-up (PACU and ward)
Measure: Mean (Standard Deviation); unit: vials
Arm/Group | Hypo | NoHypo
Number analyzed (Participants) | 37 | 41
vials
  NSAID PACU | 0.8 (0.4) | 0.96 (0.18)
  Opioid PACU | 0.1 (0.3) | 0.36 (0.49)
  NSAID ward | 2.83 (1.23) | 5.77 (1.24)
  Opioid ward | 0 (0) | 0.63 (0.71)

3. Secondary Outcome: Rescue Analgesic Time
Description: Time to first analgesic demand at gynecology ward (after transfer from PACU to gynecology ward)
Time Frame: 48 hours (time to the first analgesic demand will be recorded)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hypo | NoHypo
Number analyzed (Participants) | 37 | 41
minutes | 627 (352.89) | 203.83 (173.13)

4. Secondary Outcome: Duration of Operation
Description: the time from the the first incision to the skin to skin closure.
Time Frame: from the induction of anesthesia and the end of the surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hypo | NoHypo
Number analyzed (Participants) | 37 | 41
minutes | 115.83 (34.19) | 114.16 (34.59)

5. Secondary Outcome: Length of Hospital Stay
Description: length of hospital stay time will be recorded
Time Frame: assessed up to 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Hypo | NoHypo
Number analyzed (Participants) | 37 | 41
days | 2.66 (0.6) | 2.96 (1.32)

6. Secondary Outcome: Number of Participants With Complications Due to SHP Block
Description: intra/postoperative complications will be noted. (post-operative nausea and vomiting (PONV) or others: ie: intra-vascular local anesthetic injection, vascular puncture, hemodynamical changes after injection,.. )
Time Frame: From the SHP block time (intraoperative) until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Hypo | NoHypo
Number analyzed (Participants) | 30 | 30
Participants
  PONV | 7 | 8
  others | 0 | 0

ADVERSE EVENTS:
Time Frame: From the SHP block time (intraoperative) until discharge
Arm/Group | Hypo | NoHypo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/41
Other Adverse Events (participants affected / at risk) | 0/37 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT03428152/Prot_SAP_000.pdf